CLINICAL TRIAL: NCT05047952
Title: Randomized, Double-Blinded, Placebo-Controlled Study Evaluating Vortioxetine for Cognitive Deficits in Persons With Post-COVID-19 Condition
Brief Title: Vortioxetine for Post-COVID-19 Condition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brain and Cognition Discovery Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCDF002
Record Dates: First submitted 2021-09-12; First posted 2021-09-17 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-11

CONDITIONS: Post-COVID-19 Condition; Post-COVID-19 Syndrome; Cognitive Impairment
Keywords: vortioxetine; fatigue; long COVID; post-acute COVID syndrome PASC; long haul COVID; brain fog; cognitive deficit; cognitive dysfunction; COVID-19 sequelae; post-acute COVID-19 syndrome; Trintellix; chronic COVID syndrome; post-COVID-19 condition; long hauler; anti-inflammatory; persistent COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Cognitive Dysfunction; Fatigue; Mental Fatigue; Cognition Disorders | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vortioxetine (Experimental): Participants aged 18-64 years: start at 10 mg vortioxetine once daily for the first 2 weeks, then dosed up to 20 mg vortioxetine once daily for weeks 2-8.
  Participants aged 65+ years: start at 5 mg vortioxetine once daily for the first 2 weeks, then dosed up to 10 mg vortioxetine once daily for weeks 2-8.
  Interventions: Drug: Vortioxetine
- Placebo (Placebo Comparator): Placebo capsule taken once daily for weeks 0-8.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vortioxetine — Participants aged 18-64 years receiving vortioxetine will be provided 10 mg/day on days 1-14 of the treatment period, and will be titrated to 20 mg/day at the start of week 3 (day 15) based on study clinician judgment. For the remaining 6 weeks, the dose of vortioxetine will be 20 mg/day, unless adjudicated otherwise by a study clinician.
  Per product monograph, participants aged 65+ years receiving vortioxetine will be provided 5 mg/day on days 1-14 of the treatment period, and will be titrated to 10 mg/day at the start of week 3 (day 15) based on study clinician judgment. For the remaining 6 weeks, the dose of vortioxetine will be 10 mg/day, unless adjudicated otherwise by a study clinician.
  Arms: Vortioxetine
Drug: Placebo — A placebo pill will be taken once daily.
  Arms: Placebo

SUMMARY:
A randomized, double-blinded, placebo-controlled trial will be conducted to evaluate vortioxetine, an antidepressant with established pro-cognitive properties, for the treatment of cognitive deficits which develop during or after an infection consistent with COVID-19, continue for 2+ months, and are not explained by an alternative diagnosis (i.e., post-COVID-19 condition). Participants (aged 18-64 years) will receive vortioxetine (10-20 mg) or placebo for 8 weeks. Participants 65+ years will receive vortioxetine (5-10 mg) or placebo for 8 weeks. Changes in cognitive functioning from baseline to endpoint (week 8) will be assessed via the Digit Symbol Substitution Test (DSST). Study visits may be conducted remotely (e.g. via Zoom, by telephone), and/or in-person.

DETAILED DESCRIPTION:
A significant percentage of individuals who have recovered from acute COVID-19 infection present with unabating, non-specific, distressing, and functionally impairing symptoms (i.e., post-COVID-19 condition). Commonly reported symptoms include, but are not limited to, cognitive impairment (e.g., "brain fog"), fatigue, apathy, depression, anxiety, insomnia, anergia, and loss of appetite. Toward the aim of identifying a common nomenclature and case definition, the World Health Organization (WHO) has recently proposed the moniker 'post COVID-19 condition'. It is estimated that approximately 10-30% of persons infected with COVID-19 experience characteristic symptoms persisting for more than 12 weeks following documentation of positive COVID-19 diagnosis.

Consensus exists that the phenomenology of post-COVID-19 condition is subserved by disturbance in immune-inflammatory systems. Currently, no treatment is identified as safe and effective for post-COVID-19 condition. A candidate treatment for post-COVID-19 condition should be capable of improving measures of cognitive function (i.e., objective and subjective), motivation and energy, as well as reducing fatigue. The rationale for prioritizing cognition as a primary therapeutic target is based on a concatenation of study results reporting that cognitive complaints/deficits and fatigue are some of the most common and debilitating features of post-COVID-19 condition. Preliminary evidence suggests that some antidepressants (e.g., SSRIs) are capable of reducing respiratory complications secondary to COVID-19 via putative mechanisms including, but not limited to, sigma-1 agonism and acid sphingomyelinase.

Vortioxetine is established as pro-cognitive, as evidenced by significant improvement on both subjective and objective measures. Vortioxetine is also documented to improve anticipatory and consummatory measures of reward function/anhedonia, improve general functioning, and measures of motivation and energy. Moreover, vortioxetine is not associated with emotional blunting and has preliminary evidence of improving sleep behaviour and circadian rhythms. The candidacy of vortioxetine as an effective treatment for post-COVID-19 condition is also strengthened by evidence indicating that vortioxetine exerts modulatory effects on cellular and cytokine systems known to be activated in persons with post-COVID-19 condition. Herein, we hypothesize that vortioxetine will be more effective than placebo in the treatment of cognitive impairment in persons with post-COVID-19 condition.

ELIGIBILITY:
Inclusion Criteria

* Age 18+
* Meets WHO-defined post-COVID-19 condition (WHO definition: 'Post COVID-19 condition occurs in individuals with a history of probable or confirmed SARS-CoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis. Common symptoms include fatigue, shortness of breath, cognitive dysfunction but also others* and generally have an impact on everyday functioning. Symptoms may be new onset following initial recovery from an acute COVID-19 episode or persist from the initial illness. Symptoms may also fluctuate or relapse over time.') To ensure the above criteria is met, participants will only be included in the study if they meet all eligibility criteria more than 12 weeks from the onset of their acute Covid-19 symptoms or positive PCR/antigen test.
* Documented history of SARS-CoV-2 infection (positive PCR/antigen test during acute illness OR clinical diagnosis by physician during or after the acute illness).
* Subjective cognitive complaints as detected by the Perceived Deficits Questionnaire (PDQ)-5.
* Ability to provide written informed consent.
* Resident of Canada.

Exclusion Criteria

* Current symptoms are fully explained by major depressive disorder or bipolar disorder.
* Pre-existing conditions that may cause cognitive impairment, or symptoms similar to those seen in post-COVID-19 condition (e.g., major neurocognitive disorder, schizophrenia, chronic fatigue syndrome [CFS]/ encephalitis meningitis [EM]), as assessed by Mini International Neuropsychiatric Interview (MINI) 7.0.2.
* Inability to follow study procedures.
* Known intolerance to vortioxetine and/or prior trial of vortioxetine with demonstrated inefficacy.
* If participants are currently taking other antidepressants, they will be asked to discontinue the antidepressant for 2-4 weeks in order to participate in the study.
* Patients on other antidepressants are allowed to participate only if the antidepressant is prescribed at subtherapeutic doses for a primary indication other than mood disorders. Participants will be made aware in the consent form that the combination of the two antidepressants would be considered investigational and that the safety/efficacy profiles are unknown.
* Current alcohol or substance use disorder.
* Inability to provide consent.
* Current alcohol and/or substance use disorder as confirmed by the M.I.N.I 7.0.2.
* Presence of comorbid psychiatric disorder that is a primary focus of clinical concern as confirmed by the M.I.N.I. 7.0.2.
* Medications approved and/or employed off-label for cognitive dysfunction (e.g., psychostimulants).
* Any medication for a general medical disorder that, in the opinion of the investigator, may affect cognitive function.
* Use of benzodiazepines within 12 hours of cognitive assessments.
* Consumption of alcohol within 8 hours of cognitive assessments.
* Physical, cognitive, or language impairments sufficient to adversely affect data derived from cognitive assessments.
* Diagnosed reading disability or dyslexia.
* Clinically significant learning disorder by history.
* Electroconvulsive therapy (ECT) in the last 6 months.
* History of moderate or severe head trauma (e.g., loss of consciousness for >1 hour), other neurological disorders, or unstable systemic medical diseases that in the opinion of the investigator are likely to affect the central nervous system.
* Pregnant and/or breastfeeding.
* Received investigational agents as part of a separate study within 30 days of the screening visit.
* Actively suicidal/presence of suicidal ideation or evaluated as being at suicide risk (as per clinical judgment).
* Currently receiving treatment with Monoamine Oxidase Inhibitors (MAOIs) antidepressants, antibiotics such as linezolid, or intravenous methylene blue.
* Previous hypersensitivity reaction to vortioxetine or any components of the formulation. Angioedema has been reported in patients treated with vortioxetine.
* Serotonin syndrome.
* Abnormal bleeding.
* Previous history of mania/hypomania.
* Angle closure glaucoma.
* Hyponatremia.
* Moderate hepatic impairment.
* Active seizure disorder/epilepsy, not controlled by medication
* Presence of any unstable medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger S. McIntyre, MD, FRCPC, Principal Investigator — Brain and Cognition Discovery Foundation
Locations (1):
- Brain and Cognition Discovery Foundation (BCDF), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahase E. Covid-19: What do we know about "long covid"? BMJ. 2020 Jul 14;370:m2815. doi: 10.1136/bmj.m2815. No abstract available. PMID 32665317
- [Background] Burke MJ, Del Rio C. Long COVID has exposed medicine's blind-spot. Lancet Infect Dis. 2021 Aug;21(8):1062-1064. doi: 10.1016/S1473-3099(21)00333-9. Epub 2021 Jun 18. No abstract available. PMID 34153235
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Sudre CH, Murray B, Varsavsky T, Graham MS, Penfold RS, Bowyer RC, Pujol JC, Klaser K, Antonelli M, Canas LS, Molteni E, Modat M, Jorge Cardoso M, May A, Ganesh S, Davies R, Nguyen LH, Drew DA, Astley CM, Joshi AD, Merino J, Tsereteli N, Fall T, Gomez MF, Duncan EL, Menni C, Williams FMK, Franks PW, Chan AT, Wolf J, Ourselin S, Spector T, Steves CJ. Attributes and predictors of long COVID. Nat Med. 2021 Apr;27(4):626-631. doi: 10.1038/s41591-021-01292-y. Epub 2021 Mar 10. PMID 33692530
- [Background] Mahase E. Long covid could be four different syndromes, review suggests. BMJ. 2020 Oct 14;371:m3981. doi: 10.1136/bmj.m3981. No abstract available. PMID 33055076
- [Background] Puntmann VO, Carerj ML, Wieters I, Fahim M, Arendt C, Hoffmann J, Shchendrygina A, Escher F, Vasa-Nicotera M, Zeiher AM, Vehreschild M, Nagel E. Outcomes of Cardiovascular Magnetic Resonance Imaging in Patients Recently Recovered From Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Nov 1;5(11):1265-1273. doi: 10.1001/jamacardio.2020.3557. PMID 32730619
- [Background] Lenze EJ, Mattar C, Zorumski CF, Stevens A, Schweiger J, Nicol GE, Miller JP, Yang L, Yingling M, Avidan MS, Reiersen AM. Fluvoxamine vs Placebo and Clinical Deterioration in Outpatients With Symptomatic COVID-19: A Randomized Clinical Trial. JAMA. 2020 Dec 8;324(22):2292-2300. doi: 10.1001/jama.2020.22760. PMID 33180097
- [Background] Hoertel N, Sanchez-Rico M, Vernet R, Beeker N, Jannot AS, Neuraz A, Salamanca E, Paris N, Daniel C, Gramfort A, Lemaitre G, Bernaux M, Bellamine A, Lemogne C, Airagnes G, Burgun A, Limosin F; AP-HP / Universities / INSERM COVID-19 Research Collaboration and AP-HP COVID CDR Initiative. Association between antidepressant use and reduced risk of intubation or death in hospitalized patients with COVID-19: results from an observational study. Mol Psychiatry. 2021 Sep;26(9):5199-5212. doi: 10.1038/s41380-021-01021-4. Epub 2021 Feb 4. PMID 33536545
- [Background] Christensen MC, Loft H, McIntyre RS. Vortioxetine improves symptomatic and functional outcomes in major depressive disorder: A novel dual outcome measure in depressive disorders. J Affect Disord. 2018 Feb;227:787-794. doi: 10.1016/j.jad.2017.11.081. Epub 2017 Nov 16. PMID 29689693
- [Background] McIntyre RS, Florea I, Tonnoir B, Loft H, Lam RW, Christensen MC. Efficacy of Vortioxetine on Cognitive Functioning in Working Patients With Major Depressive Disorder. J Clin Psychiatry. 2017 Jan;78(1):115-121. doi: 10.4088/JCP.16m10744. PMID 27780334
- [Background] McIntyre RS, Harrison J, Loft H, Jacobson W, Olsen CK. The Effects of Vortioxetine on Cognitive Function in Patients with Major Depressive Disorder: A Meta-Analysis of Three Randomized Controlled Trials. Int J Neuropsychopharmacol. 2016 Jun 15;19(10):pyw055. doi: 10.1093/ijnp/pyw055. PMID 27312740
- [Background] Cao B, Park C, Subramaniapillai M, Lee Y, Iacobucci M, Mansur RB, Zuckerman H, Phan L, McIntyre RS. The Efficacy of Vortioxetine on Anhedonia in Patients With Major Depressive Disorder. Front Psychiatry. 2019 Jan 31;10:17. doi: 10.3389/fpsyt.2019.00017. eCollection 2019. PMID 30766492
- [Background] Subramaniapillai M, Mansur RB, Zuckerman H, Park C, Lee Y, Iacobucci M, Cao B, Ho R, Lin K, Phan L, McIntyre RS. Association between cognitive function and performance on effort based decision making in patients with major depressive disorder treated with Vortioxetine. Compr Psychiatry. 2019 Oct;94:152113. doi: 10.1016/j.comppsych.2019.07.006. Epub 2019 Jul 24. PMID 31404802
- [Background] Fagiolini A, Florea I, Loft H, Christensen MC. Effectiveness of Vortioxetine on Emotional Blunting in Patients with Major Depressive Disorder with inadequate response to SSRI/SNRI treatment. J Affect Disord. 2021 Mar 15;283:472-479. doi: 10.1016/j.jad.2020.11.106. Epub 2020 Nov 19. PMID 33516560
- [Background] Cao B, Park C, Rosenblat JD, Chen Y, Iacobucci M, Subramaniapillai M, Mansur RB, Zuckerman H, Lee Y, McIntyre RS. Changes in sleep predict changes in depressive symptoms in depressed subjects receiving vortioxetine: An open-label clinical trial. J Psychopharmacol. 2019 Nov;33(11):1388-1394. doi: 10.1177/0269881119874485. Epub 2019 Sep 18. PMID 31530216
- [Background] Talmon M, Rossi S, Pastore A, Cattaneo CI, Brunelleschi S, Fresu LG. Vortioxetine exerts anti-inflammatory and immunomodulatory effects on human monocytes/macrophages. Br J Pharmacol. 2018 Jan;175(1):113-124. doi: 10.1111/bph.14074. Epub 2017 Nov 28. PMID 29057467
- [Background] Tomaz VS, Chaves Filho AJM, Cordeiro RC, Juca PM, Soares MVR, Barroso PN, Cristino LMF, Jiang W, Teixeira AL, de Lucena DF, Macedo DS. Antidepressants of different classes cause distinct behavioral and brain pro- and anti-inflammatory changes in mice submitted to an inflammatory model of depression. J Affect Disord. 2020 May 1;268:188-200. doi: 10.1016/j.jad.2020.03.022. Epub 2020 Mar 6. PMID 32174477
- [Background] Mahableshwarkar AR, Zajecka J, Jacobson W, Chen Y, Keefe RS. A Randomized, Placebo-Controlled, Active-Reference, Double-Blind, Flexible-Dose Study of the Efficacy of Vortioxetine on Cognitive Function in Major Depressive Disorder. Neuropsychopharmacology. 2015 Jul;40(8):2025-37. doi: 10.1038/npp.2015.52. Epub 2015 Feb 17. PMID 25687662
- [Background] Ceban F, Ling S, Lui LMW, Lee Y, Gill H, Teopiz KM, Rodrigues NB, Subramaniapillai M, Di Vincenzo JD, Cao B, Lin K, Mansur RB, Ho RC, Rosenblat JD, Miskowiak KW, Vinberg M, Maletic V, McIntyre RS. Fatigue and cognitive impairment in Post-COVID-19 Syndrome: A systematic review and meta-analysis. Brain Behav Immun. 2022 Mar;101:93-135. doi: 10.1016/j.bbi.2021.12.020. Epub 2021 Dec 29. PMID 34973396
- [Background] Soriano JB, Murthy S, Marshall JC, Relan P, Diaz JV; WHO Clinical Case Definition Working Group on Post-COVID-19 Condition. A clinical case definition of post-COVID-19 condition by a Delphi consensus. Lancet Infect Dis. 2022 Apr;22(4):e102-e107. doi: 10.1016/S1473-3099(21)00703-9. Epub 2021 Dec 21. PMID 34951953
- [Background] Davis HE, Assaf GS, McCorkell L, Wei H, Low RJ, Re'em Y, Redfield S, Austin JP, Akrami A. Characterizing long COVID in an international cohort: 7 months of symptoms and their impact. EClinicalMedicine. 2021 Aug;38:101019. doi: 10.1016/j.eclinm.2021.101019. Epub 2021 Jul 15. PMID 34308300
- [Derived] Liao S, Teopiz KM, Kwan ATH, Le GH, Wong S, Ballum H, Rhee TG, Badulescu S, Cao B, Guo Z, Meshkat S, Phan L, Subramaniapillai M, Ho R, McIntyre RS. Relationship between anhedonia and psychosocial functioning in post-COVID-19 condition: a post-hoc analysis. Curr Med Res Opin. 2024 Aug;40(8):1407-1411. doi: 10.1080/03007995.2024.2374510. Epub 2024 Jul 8. PMID 38954402
- [Derived] Teopiz KM, Kwan ATH, Le GH, Guo Z, Badulescu S, Ceban F, Meshkat S, Di Vincenzo JD, d'Andrea G, Cao B, Ho R, Rhee TG, Dev DA, Phan L, Subramaniapillai M, Mansur RB, Rosenblat JD, McIntyre RS. Association between fatigue and depressive symptoms in persons with post-COVID-19 condition: a post hoc analysis. Curr Med Res Opin. 2024 Jul;40(7):1203-1209. doi: 10.1080/03007995.2024.2360647. Epub 2024 Jun 11. PMID 38860901
- [Derived] Kwan ATH, Guo Z, Ceban F, Le GH, Wong S, Teopiz KM, Rhee TG, Ho R, Di Vincenzo JD, Badulescu S, Meshkat S, Cao B, Rosenblat JD, d'Andrea G, Dev DA, Phan L, Subramaniapillai M, McIntyre RS. Assessing the Effects of Metabolic Disruption, Body Mass Index and Inflammation on Depressive Symptoms in Post-COVID-19 Condition: A Randomized Controlled Trial on Vortioxetine. Adv Ther. 2024 May;41(5):1983-1994. doi: 10.1007/s12325-024-02826-9. Epub 2024 Mar 23. PMID 38520501
- [Derived] Kwan ATH, Le GH, Guo Z, Ceban F, Teopiz KM, Rhee TG, Ho R, Di Vincenzo JD, Badulescu S, Meshkat S, Cao B, Rosenblat JD, Dev DA, Phan L, Subramaniapillai M, McIntyre RS. Impacts of metabolic disruption, body mass index and inflammation on cognitive function in post-COVID-19 condition: a randomized controlled trial on vortioxetine. Ann Gen Psychiatry. 2024 Feb 29;23(1):10. doi: 10.1186/s12991-024-00494-1. PMID 38424537
- [Derived] Le GH, Kwan ATH, Wong S, Guo Z, Teopiz KM, Badulescu S, Meshkat S, d'Andrea G, Ho R, Rhee TG, Cao B, Phan L, Rosenblat JD, Mansur RB, Subramaniapillai M, McIntyre RS. Impact of Elevated Body Mass Index (BMI) on Hedonic Tone in Persons with Post-COVID-19 Condition: A Secondary Analysis. Adv Ther. 2024 Feb;41(2):686-695. doi: 10.1007/s12325-023-02760-2. Epub 2023 Dec 19. PMID 38114867
- See also: World Health Organization (WHO) COVID-19 Dashboard — https://covid19.who.int
- See also: An Analysis of the Prolonged COVID-19 Symptoms Survey by Patient-Led Research Team — https://patientresearchcovid19.com/research/report-1/
- See also: Study With Vortioxetine on Emotional Functioning in Patients With Depression (COMPLETE) — https://clinicaltrials.gov/ct2/show/NCT03835715

RESULTS

PARTICIPANT FLOW:
Groups:
- Vortioxetine: Participants aged 18-64 years: start at 10 mg vortioxetine once daily for the first 2 weeks, then dosed up to 20 mg vortioxetine once daily for weeks 2-8.
  Participants aged 65+ years: start at 5 mg vortioxetine once daily for the first 2 weeks, then dosed up to 10 mg vortioxetine once daily for weeks 2-8.
  Vortioxetine: Participants aged 18-64 years receiving vortioxetine will be provided 10 mg/day on days 1-14 of the treatment period, and will be titrated to 20 mg/day at the start of week 3 (day 15) based on study clinician judgment. For the remaining 6 weeks, the dose of vortioxetine will be 20 mg/day, unless adjudicated otherwise by a study clinician.
  Per product monograph, participants aged 65+ years receiving vortioxetine will be provided 5 mg/day on days 1-14 of the treatment period, and will be titrated to 10 mg/day at the start of week 3 (day 15) based on study clinician judgment. For the remaining 6 weeks, the dose of vortioxetine will be 10 mg/day, unless adjudicated otherwise by a study clinician.
Period: Overall Study
Arm/Group | Vortioxetine | Placebo
Started | 75 | 74
Completed | 68 | 73
Not Completed | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vortioxetine | Placebo | Total
Number analyzed (Participants) | 75 | 74 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.65 (12.26) | 44.94 (12.03) | 44.36 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 47 | 98
  Male | 24 | 27 | 51
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 58 | 55 | 113
  Non-Caucasian | 17 | 19 | 36
Region of Enrollment [Number; unit: participants]
  Canada | 75 | 74 | 149
Confirmed COVID Diagnosis [Number; unit: participants] | 59 | 59 | 118
Lifetime Major Depressive Disorder Diagnosis [Number; unit: participants] | 32 | 25 | 57
Highest Education = Highschool [Number; unit: participants] | 18 | 14 | 32
Highest Education = College/University [Number; unit: participants] | 47 | 42 | 89
Highest Education - Graduate School [Number; unit: participants] | 10 | 18 | 28
Combined Digit Symbol Substitution Test [Mean (Standard Deviation); unit: units on a scale] — The combined Z-score for the Digit Symbol Substitution Test (DSST) represents a standardized measure of the overall performance or outcome both the computerized DSST and the paper-based DSST. Positive Z-scores might suggest above-average performance, Z-score of 0 represents the mean performance, while negative Z-scores suggest below-average performance.
  units on a scale | -0.02 (0.91) | -0.21 (0.96) | -0.07127 (1.002)
Computurized Digit Symbol Substitution Test (DSST) [Mean (Standard Deviation); unit: Total Number of Symbols] — The Computerized DSST is the DSST that has been converted to an online version that can be done remotely. This score represents only the score from the Computerized DSST. The score ranges are from 18-84, with higher scores representing better outcome on the task.
  Total Number of Symbols | 48.40 (10.11) | 46.35 (10.75) | 47.36 (10.50)
Remote Participation in Trial, n (%) [Number; unit: participants] | 38 | 40 | 78
The Quick Inventory of Depressive Symptomatology-Self-report (QIDS-SR16) [Mean (Standard Deviation); unit: Total Score] — The Quick Inventory of Depressive Symptomatology (QIDS-SR16) measures the subjective severity of depressive symptoms. Total Score is reported (total range=0-27) with higher scores being associated with increased severity in depressive symptoms. Lower scores are associated with decreased severity in depressive symptoms.
  Total Score | 10.03 (4.33) | 10.32 (4.37) | 10.18 (4.33)
The 5-item World Health Organization Well-Being Index (WHO-5) [Mean (Standard Deviation); unit: Total Score] — The (WHO-5 is a self-report instrument measuring mental well-being. The total score ranges from zero to 25, zero representing worst possible mental well-being and 25 representing best possible mental well-being.
  Total Score | 9.808 (4.579) | 9.757 (9.808) | 9.808 (4.245)

OUTCOME MEASURES:

1. Primary Outcome: Least Square Mean Change in Baseline to Week 8 on Z-score in Combined Digit Symbol Substitution Test (DSST)
Description: This measures the least square mean change in baseline-to-end point on z-score on the combined DSST. Depicted is the least square (LS) mean [standard error of mean (SEM)] change in DSST z-scores from baseline to week 8 using an independent covariance matrix with time as a categorical variable, adjusted for the type of cognitive test (Pen/Paper versus Online CogState version). Larger least squares mean indicates a higher predicted or adjusted average outcome for that group or condition compared to others. In other words, if you have a higher least squares mean for a treatment group, it suggests that, after adjusting for the effects of other variables, that group tends to have a higher average outcome, indicating better performance. A least squares mean of 0 indicates that the groups has no difference in average outcome. There is no fixed maximum or minimum for LS Means. They are derived from the data and can, in principle, take any real value (positive, negative, or zero)
Time Frame: Weeks 0-8
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vortioxetine | Placebo
Number analyzed (Participants) | 75 | 74
score on a scale | 0.332 (0.0752) | 0.184 (0.0934)

2. Secondary Outcome: Baseline to Endpoint Change in World Health Organization Wellbeing Scale, 5-item (WHO-5)
Description: This measures the least square mean change in baseline-to-end point on scores on the WHO-5. Depicted is the least square (LS) mean [standard error of mean (SEM)] change in WHO-5 from baseline to week 8. Larger least squares mean indicates a higher predicted or adjusted average outcome for that group or condition compared to others. In other words, if you have a higher least squares mean for a treatment group, it suggests that, after adjusting for the effects of other variables, that group tends to have a higher average outcome, indicating better performance. A least squares mean of 0 indicates that the groups has no difference in average outcome. There is no fixed maximum or minimum for LS Means. They are derived from the data and can, in principle, take any real value (positive, negative, or zero)
Time Frame: Weeks 0-8
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vortioxetine | Placebo
Number analyzed (Participants) | 67 | 73
score on a scale | 1.759 (0.489) | 1.107 (0.590)

3. Secondary Outcome: Baseline-to-endpoint (i.e., Week 8) Change in the Quick Inventory of Depressive Symptomology, Self Report (QIDS-SR-16)
Description: This measures the least square mean change in baseline-to-end point on the QIDS-SR-16. A negative least squares estimate for the QIDS-SR-16 score from baseline to week 8 indicates a reduction in depressive symptoms. Specifically, it implies that, on average, the QIDS-SR-16 scores have decreased over the 8-week period. Since lower QIDS-SR-16 scores correspond to less severe depressive symptoms, a negative change is a positive outcome, showing improvement. A least squares mean of 0 indicates that the groups has no difference in average outcome. There is no fixed maximum or minimum for LS Means. They are derived from the data and can, in principle, take any real value (positive, negative, or zero)
Time Frame: Week 0-8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vortioxetine | Placebo
Number analyzed (Participants) | 67 | 73
units on a scale | -3.351 (0.524) | -1.756 (0.503)

ADVERSE EVENTS:
Time Frame: Adverse events will be collected from baseline (Week 1) to endpoint (Week 8).
Arm/Group | Vortioxetine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/74
Other Adverse Events (participants affected / at risk) | 47/75 | 34/74
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vortioxetine (N=75) | Placebo (N=74)
Fatigue (Nervous system disorders) | 8 (8) | 8 (8)
Nausea (Gastrointestinal disorders) | 36 (36) | 19 (19)
Headache (Nervous system disorders) | 6 (6) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 11 (11)
Constipation (Gastrointestinal disorders) | 7 (7) | 2 (2)
Dyspepsia (Cardiac disorders) | 6 (6) | 8 (8)

LIMITATIONS AND CAVEATS:
participants not stratified as part of eligibility on the basis of having a predetermined threshold of objective cognitive impairment prior to enrolment. Participants in our study were primarily recruited via media announcements including presentations at Post COVID-19 Condition online groups. Our sample was not recruited from a medical clinic including "Post COVID-19 Condition clinics." Majority of participants were Caucasian; it is recognized that our results may not generalizable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT05047952/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT05047952/ICF_001.pdf